CLINICAL TRIAL: NCT00979771
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Investigate the Ability of GSK706769 to Maintain Clinical Remission After Withdrawal of Enbrel in Patients With Rheumatoid Arthritis
Brief Title: A Study to Investigate the Ability of GSK706769 to Maintain Clinical Remission After Withdrawal of Enbrel in Rheumatoid Arthritis Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Cancelled Before Active
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 112145; 2009-012204-42 (EudraCT Number)
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Arthritis, Rheumatoid
Keywords: GSK706769; Enbrel; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK706769 (Experimental): 100 mg GSK706769 twice daily orally (BID) for 28 days
  Interventions: Drug: GSK706769
- Placebo (Placebo Comparator): GSK706769 matched-placebo twice daily orally (BID) for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK706769 — 100 mg GSK706769 twice daily orally (BID) for 28 days
  Arms: GSK706769
Drug: Placebo — GSK706769 matched-placebo twice daily orally (BID) for 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if GSK706769 can maintain clinical remission established by Enbrel after withdrawal of Enbrel in rheumatoid arthritis patients.

DETAILED DESCRIPTION:
This study is a phase II, randomized, double-blind, placebo-controlled, parallel group study in subjects with rheumatoid arthritis (RA) on stable doses of Enbrel. Subjects with an adequate response to Enbrel will be enrolled into the study. Subjects will be withdrawn from their Enbrel and randomized to receive 28 days of dosing with either GSK706769 or placebo followed by 28 days off-drug. This study is exploring a novel therapeutic paradigm for RA, remission maintenance. In such an approach, remission is induced and then the inducing agent is stopped and a maintenance agent is added. The clinical benefit would be derived from the fact that the remission agent may be easier to take (e.g. oral rather than parenteral), more durable in its maintenance of remission, and/or safer (e.g. no TB reactivation). This study directly explores remission maintenance. Specifically, in a randomised, double blind, placebo controlled study, RA patients in remission through an adequate response to Enbrel will be recruited. Enbrel has been selected as it has a relatively short half life and therefore it is more likely patients treated with placebo may have a higher incidence of relapse after 28 days than with other anti-TNF treatments. After withdrawal of Enbrel (and possibly other oral DMARDs), subjects will be randomised to receive GSK706769 or placebo for 28 days followed by a period of 28 days off treatment. It is hypothesized that GSK706769 will prevent any CCR5+ cells from returning into the synovium, thereby resulting in maintenance of the efficacy induced by Enbrel. In the placebo group, CCR5 cells may re-populate the synovium resulting in increased inflammation. Patients experiencing increased disease activity will be able to withdraw from the study and resume standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time Female subjects must agree to use contraception until 4 days post-last dose.
* Body weight greater than or equal to 50 kg and BMI within the range 19 - 32 kg/m2.
* The subject has a diagnosis of RA according to the revised 1987 criteria of the American College of Rheumatology (ACR) and has been treated with an anti TNF-alpha agent for < 2 years.
* The subject is taking Enbrel for at least 6 months prior to enrollment.
* The subject is willing to stop taking Enbrel for 56 days.
* The subject is in clinical remission, defined as DAS28 less than or equal to 2.6 and has been for the preceding 6 months.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
* AST and ALT < 2xULN; alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* The subject is using oral prednisolone at doses > 10mg/day.
* The subject's NSAID or glucocorticoid dosing regimen has changed during the 4 weeks prior to randomisation.
* The subject's receiving DMARDs other than Enbrel and methotrexate.
* The subject's current methotrexate regimen has changed significantly (i.e. likely to impact disease activity during the study period) within the 3 months prior to dosing e.g. changes in dose of greater than 2.5mg.
* Use of CYP3A4 inhibitors/inducers within 14 days prior to dosing and CYP3A4 substrates with a narrow therapeutic index within 7 days prior to dosing.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Absolute neutrophil count < 1500/ul.
* History of sensitivity to the study medication, or components thereof or a history of drug or other allergy that contraindicates their participation.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug screen, unless the subject is receiving a prescribed medication that could give a positive in the drug screen and prior to the screen being sent the medication has been discussed and pre-approved by the medical monitor.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined by the protocol.
* The subject has an acute infection or a history of repeated or chronic infections.
* The subject has significant cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions that in the opinion of the investigator and/or medical monitor, places the subject at an unacceptable risk as a participant in this trial.
* Subjects with autoimmune hemolytic anemia or G6PD deficiency.
* Malignancy in the past 2 years, except for adequately treated non-invasive cancers of the skin.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Consumption of grapefruit, grapefruit juice or grapefruit hybrids within 7 days prior to the first dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02-01 (Estimated); Primary Completion 2011-04-28 (Estimated); Study Completion 2011-04-28 (Estimated)

PRIMARY OUTCOMES:
Maintenance of clinical remission after withdrawal of Enbrel in patients with RA, as determined by DAS28 scores. | Day 28 after first dose administration

SECONDARY OUTCOMES:
The ability of GSK706769 to maintain clinical remission after withdrawal of Enbrel in patients with RA, as determined by the Patient Global Assessment scores and evidence of swollen or tender joints. | Day 28 and 28 days after last dose of study medication
To investigate the time to relapse following withdrawal of Enbrel | After first dose administration
Safety and tolerability of GSK706769 following repeat dosing in RA subjects for up to 28 days | After first dose administration
Rheumatological assessments, pain, fatigue and physical functioning following repeat dosing with GSK706769 for up to 28 days | Day 1, 14, 28, 56 after first dose administration
Pharmacokinetics (PK) of GSK706769, and its metabolite GSK1996847A | Day 1, 14 and 28 after first dose administration
CCR5 receptor occupancy (RO) in peripheral blood following repeat dosing with GSK706769 for up to 28 days, as feasible | Day 1, 14 and 28 after first dose administration

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Amsterdam, Netherlands